CLINICAL TRIAL: NCT00022386
Title: An Open-Label Study of PROCRIT (Epoetin Alfa) in Women Undergoing Adjuvant Chemotherapy for Stage I, II, or III Breast Cancer
Brief Title: Epoetin Alfa in Treating Chemotherapy-Related Anemia in Women With Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: ORTHO-PR-00-27-012; UCLA-0011004; CDR0000068811 (Registry Identifier: PDQ (Physician Data Query)); ORTHO-PR-01-27-003; NCI-G01-2002
Record Dates: First submitted 2001-08-10; First posted 2004-04-05 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2002-05

CONDITIONS: Anemia; Breast Cancer; Fatigue
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; anemia; fatigue
MeSH Terms: conditions — Anemia; Breast Neoplasms; Fatigue | interventions — Epoetin Alfa

INTERVENTIONS:
Biological: epoetin alfa
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Epoetin alfa may stimulate red blood cell production to treat patients who have anemia following chemotherapy.

PURPOSE: Phase IV trial to study the effectiveness of epoetin alfa in treating chemotherapy-related anemia in women who have stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effectiveness and safety of epoetin alfa in patients receiving adjuvant chemotherapy for stage I, II, or III breast cancer. II. Determine the clinical outcomes in these patients receiving this drug.

OUTLINE: This is a multicenter study. Patients receive epoetin alfa subcutaneously once weekly for up to 24 weeks in the absence of unacceptable toxicity. Quality of life is assessed at baseline, at week 13, and at study completion.

PROJECTED ACCRUAL: A maximum of 2,500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage I, II, or III breast cancer Planned adjuvant anthracycline-based chemotherapy with or without a taxane for 3-6 months Hemoglobin 10-14 g/dL (independent of transfusion) No anemia due to factors other than cancer/chemotherapy (i.e., iron, cyanocobalamin, or folate deficiency; hemolysis; gastrointestinal bleeding; or myelodysplastic syndrome) Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: At least 9 months Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified Cardiovascular: No uncontrolled or severe cardiovascular disease No myocardial infarction within the past 6 months No uncontrolled hypertension No congestive heart failure Other: No hypersensitivity to mammalian cell-derived products No hypersensitivity to human albumin Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 months since prior epoetin alfa or any investigational forms of erythropoietin (e.g., gene-activated erythropoietin or novel erythropoiesis- stimulating protein) No transfusion within the past 30 days No other concurrent epoetin alfa Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No other concurrent investigational drugs No other concurrent treatments for anemia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A. Glaspy, MD, MPH, Study Chair — Jonsson Comprehensive Cancer Center